CLINICAL TRIAL: NCT05872997
Title: Effectiveness of Mobilization With Movement Along With Sensory Motor Training in Patients With Knee Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: DPT/Batch-Fall18/537
Record Dates: First submitted 2023-03-18; First posted 2023-05-24 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mobilization With Movement (Experimental): Mobilization With Movement
  Interventions: Diagnostic Test: Sensory Motor Training

INTERVENTIONS:
Diagnostic Test: Sensory Motor Training — Mobilization With Movement Along With Sensory Motor Training

SUMMARY:
to find out the Effectiveness of Mobilization With Movement Along With Sensory Motor Training in Patients With Knee Osteoarthritis

ELIGIBILITY:
Inclusion Criteria:

* Both genders between age of 45 and 70 with knee pain more than 3 months of presentation in outpatient department. They were also required to stand independently from sitting and prone lying

Exclusion Criteria:

* Patients with any lower limb fractures, any neurological condition, contraindication to manual therapy, post traumatic Knee osteoarthritis, total knee replacement, uncontrolled hypertension, and radiating leg pain

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-05-30 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Oxford Scale | 6 Months
  Effectiveness of Mobilization With Movement Along With Sensory Motor Training using Oxford Scale
Numeric Pain Scale | 6 Months
  Effectiveness of Mobilization With Movement Along With Sensory Motor Training using Numeric Pain Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Chaudary Muhammad Akram Teaching Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No